CLINICAL TRIAL: NCT07106099
Title: Effectiveness of The Diagnostic Training on The Signs and Rısks of Child Abuse and Neglect Given By The Tell-What You Have Learned Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Associate Professor Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SBÜ-AYDINKARTAL-009
Record Dates: First submitted 2024-12-08; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-01

CONDITIONS: Child Abuse; Neglect
Keywords: Midwifery; Child Abuse; Child Neglect; Student; Teach-Back Method

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (n:43) (No Intervention): Students in the control group will be given 2 hours of training on diagnosing the symptoms and risks of child abuse and neglect using the classical method.
- intervention group (n:43) (Experimental): Students in the intervention group will be given training on identifying the symptoms and risks of child abuse and neglect using the tell-what-you-learned method.
  Interventions: Behavioral: Training given with the tell-what-you-learned method

INTERVENTIONS:
Behavioral: Training given with the tell-what-you-learned method — Students in the intervention group will be given training on diagnosing the symptoms and risks of child abuse and neglect, given by the tell-what-you-learned method, and will be given a practice in which its effectiveness will be evaluated.
  Arms: intervention group (n:43)

SUMMARY:
The research, planned in an experimental design with a pretest-posttest control group, was conducted with second-year students studying at the Department of Midwifery (n=86). The students participating in the study were divided into intervention (n: 43) and control (n: 43) groups by simple random sampling. Training in identifying the symptoms and risks of child abuse and neglect was given to the intervention group students with the explain method, while the control group was given classical training. In collecting data; 'Introductory Information Form', 'Identification Scale for Symptoms and Risks of Child Abuse and Neglect', and 'Child Abuse and Neglect Awareness Scale' were used. Data were collected before the application and at the 4th week after the application.

DETAILED DESCRIPTION:
The implementation phase of the research was carried out in the classroom of the Midwifery Department at the Faculty of Health Sciences of a public university. During the training sessions, all student activities were observed by the researchers.

Second-year midwifery students (n=86) were randomly assigned by the researchers to the intervention group (n=43) and the control group (n=43) using the website https://www.randomizer.org/. An introductory information form was administered to all participants, and a briefing session was held before the implementation. In this session, detailed information about the procedures to be carried out in the study was provided, and a question-and-answer session was conducted. Students were informed about the training plan's flowchart, content, process, and environment. It was explained that the intervention group (n=43) would be trained on identifying signs and risks of child abuse and neglect using the "teach-back method," while the control group (n=43) would receive traditional education on the same topic.

Before the training, as a pretest, the "Scale for Identifying Signs and Risks of Child Abuse and Neglect" and the "Child Abuse and Neglect Awareness Scale" were administered to all participants. All groups were given a 2-hour theoretical session on child abuse and neglect via a PowerPoint presentation. During the session, students' questions were addressed. At the end of the training, all students were asked to leave the classroom. Subsequently, intervention group students were brought back individually and asked to explain the training content in their own words. After their explanations, they were asked additional questions such as "Is there anything you would like to add?" and "Can you provide examples related to the topic?" to encourage further elaboration.

Four weeks after the training, all participants were administered the same scales as a posttest: the "Scale for Identifying Signs and Risks of Child Abuse and Neglect" and the "Child Abuse and Neglect Awareness Scale."

ELIGIBILITY:
Inclusion Criteria:

* Being a second-year student at the University of Health Sciences, Hamidiye Faculty of Health Sciences, Department of Midwifery
* Volunteering to participate in research

Exclusion Criteria:

* Students who do not meet the sample selection criteria
* Not being willing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
introductory information form | Baseline
  The survey form prepared by the researchers based on the literature consists of two parts. In the first section, there are questions about socio-demographic information (age, gender, marital status, educational status, family type). In the second part, there are questions assessing their knowledge and attitudes about child abuse and neglect.
Scale for Identification of Symptoms and Risks of Child Abuse and Neglect | through study completion, an average of 1 year
  There are 6 subscales of the scale form (ÇİİBRTÖ) for diagnosing the symptoms and risks of child abuse and neglect developed by Uysal. It is a Likert-type scale consisting of 67 items to determine the knowledge levels of nurses and midwives in diagnosing the symptoms and risks of child abuse and neglect. The answers given to the questions in the scale vary between 1 and 5 points. A high mean score from the sub-dimensions of the scale means that the level of knowledge in that field is high. The highest score that can be obtained from the scale is 335 and the lowest score is 67.
Child Abuse and Neglect Awareness Scale | through study completion, an average of 1 year
  The scale was developed for the first time in 2014 as part of the thesis study, and its validity and reliability studies were conducted. Child abuse and neglect awareness scale (ÇİİFÖ) consists of 20 items, 11 of which are negative and 9 of which are positive, which can be grouped under 4 subgroups (physical abuse, sexual abuse, emotional abuse and neglect). It is a 5-point Likert type scale (ranging from 1 to 5, between "definitely not suitable" and "definitely suitable"). The highest score to be obtained from the scale is 100 and the lowest score is 20. As the scores obtained from the scale increase, the level of awareness of child abuse and neglect increases, and as the scores decrease, the level of awareness of child abuse and neglect decreases. Its reliability was determined by internal consistency and test-retest methods. In the study, the Cronbach's Alpha value of the scale was found to be 0.76.

SECONDARY OUTCOMES:
Scale for Identification of Symptoms and Risks of Child Abuse and Neglect | through study completion, an average of 1 year
  There are 6 subscales of the scale form (ÇİİBRTÖ) for diagnosing the symptoms and risks of child abuse and neglect developed by Uysal. It is a Likert-type scale consisting of 67 items to determine the knowledge levels of nurses and midwives in diagnosing the symptoms and risks of child abuse and neglect. The answers given to the questions in the scale vary between 1 and 5 points. A high mean score from the sub-dimensions of the scale means that the level of knowledge in that field is high. The highest score that can be obtained from the scale is 335 and the lowest score is 67.
Child Abuse and Neglect Awareness Scale | through study completion, an average of 1 year
  The scale was developed for the first time in 2014 as part of the thesis study, and its validity and reliability studies were conducted. Child abuse and neglect awareness scale (ÇİİFÖ) consists of 20 items, 11 of which are negative and 9 of which are positive, which can be grouped under 4 subgroups (physical abuse, sexual abuse, emotional abuse and neglect). It is a 5-point Likert type scale (ranging from 1 to 5, between "definitely not suitable" and "definitely suitable"). The highest score to be obtained from the scale is 100 and the lowest score is 20. As the scores obtained from the scale increase, the level of awareness of child abuse and neglect increases, and as the scores decrease, the level of awareness of child abuse and neglect decreases. Its reliability was determined by internal consistency and test-retest methods. In the study, the Cronbach's Alpha value of the scale was found to be 0.76.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin AYDIN KARTAL, Doç. Dr., Principal Investigator — yasemin.aydin@sbu.edu.tr; Büşra HIZLIOL, Arş. Gör., Study Chair — busra.hizliol@sbu.edu.tr
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No